CLINICAL TRIAL: NCT04007757
Title: Recovery and Outcomes From Stroke (ROSE) Sub-study of Genetic and Environmental Risk Factors for Hemorrhagic Stroke
Brief Title: Recovery and Outcomes From Stroke
Acronym: ROSE
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Massachusetts General Hospital (Other); University of Maryland, Baltimore (Other); Duke University, Durham, NC (Unknown); Columbia University (Other); University of Illinois at Chicago (Other); Baptist Health, Louisville (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Daniel Woo, M.D.,Professor, State University of New York at Buffalo
Other Study IDs: R01NS100417 (NIH); R01NS100417 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-07-05 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Hemorrhagic Stroke; Intracerebral Hematoma
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, DNA, RNA and complete blood count (CBC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants who have had a hemorrhagic stroke and have been enrolled into the Genetic and Environmental Risk Factors for Hemorrhagic Stroke Study who live in the area of University of Cincinnati, Massachusetts General Hospital, University of Maryland, Duke University, Columbia University and University of Chicago Illinois, age 18 years or greater. Ability of participant or legal representative to provide informed consent. Racial/ethnic category of Caucasian, African American or Hispanic.

SUMMARY:
The investigators will perform follow-up on 500 cases of deep and lobar intracerebral hemorrhage to perform advanced neuroimaging before 45 days post stroke, and evaluations of motor and cognitive function at baseline, 3 months and 6 months to determine predictors of recovery, progressive cognitive or functional impairment.

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and the leading cause of adult disability in the United States. More adults are affected by stroke each year than Alzheimer's disease, multiple sclerosis, amyotrophic lateral sclerosis or Parkinson's disease. Hemorrhagic strokes represent the most severe subtypes of stroke. An estimated 40-50% of hemorrhagic stroke victims will die and more than 80% of survivors remain disabled after hemorrhagic stroke. Yet the vast majority of analyses on outcome after stroke have focused principally on gross measures of functional outcome.

Furthermore hemorrhagic stroke differs from ischemic stroke where a loss of blood causes the area affected to be readily visible on scanning. But with hemorrhagic stroke, not only the area that we can directly see, but nearby tracts that have been compressed or stretched by the mass of the hemorrhage can be injured.

The investigators propose to follow-up on 500 cases of deep and lobar ICH to perform serial evaluations of motor and cognitive function and advanced neuroimaging to determine predictors of recovery, progressive cognitive or functional impairment. Our proposal has the advantages of adding onto a prospective ICH study which will identify and recruit cases, ability to evaluate for the degree and impact of survival and severity biases, baseline neuroimaging which includes baseline MRI, biologic samples including genotyping for apolipoprotein E alleles and uniform phenotype definitions as well as expertise in recovery/outcome analyses, advanced neuroimaging processes and epidemiologic study. This proposal performs detailed cognitive, motor and functional assessments on cases of intracerebral hemorrhage and correlates with tractography imaging. The investigators hypothesize that unlike ischemic stroke, the mass effect of the hemorrhage itself may disrupt nearby tracts in some patients while preserving them in others and will serve as a better predictor of who may recover after ICH. This project will represent the largest number of ICH cases in which tractography imaging has been performed to date.

Specific Aim #1: Improve motor recovery prediction after supratentorial ICH by adding proportion of tract injury as measured by diffusion tensor imaging (DTI) independent of the ICH volume, location, age, gender and intraventricular hemorrhage (IVH).

Hypothesis #1a: Increasing severity of injury to corticospinal tracts in ICH patients will predict worse specific motor deficits assessed at 3-month and 6-month post-stroke.

Hypothesis #1b. Injury to cortical-cortical tracts including the superior longitudinal fasciculus, uncinate fasciculus, cingulum, and arcuate fasciculus, will predict greater impairment in corresponding cognitive domains including attention, memory, executive function, and language function assessed at 3 and 6-month post-stroke.

Specific Aim #2: Determine the association of periventricular tract injury in intraventricular hemorrhage complicating ICH with subsequent incontinence and gait ataxia.

Hypothesis #2: Patients with IVH will be associated with greater periventricular tract injury than patients without IVH and that this injury will be independently associated with long-term neurogenic incontinence and gait instability after controlling for severity of the ICH including location and volume, age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater, fulfillment of the criteria for Deep, Subcortical or Lobar Intracerebral Hemorrhage (ICH)
* No evidence of trauma, vascular malformation or aneurysm, or brain tumor as a cause of ICH.
* Ability of the patient or legal representative to provide informed consent

Exclusion Criteria:

* Brainstem or Cerebellar ICH
* Patients Severely Affected by the ICH, Early Mortality, Hospice, or Withdraw of Care NOT eligible for ROSE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants already enrolled in Genetic and Environmental Risk Factors for Hemorrhagic Stroke
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change motor recovery prediction after supratentorial intracerebral hemorrhage(ICH) | Ongoing/completed end of August 2020
  This measure will determined by adding proportion of tract injury as measured by diffusion tensor imaging(DTI) methods. Measures are independent of the presenting Glasgow Coma Scale(GCS),ICH volume,location,age,sex and intraventricular hemorrhage (IVH).The primary outcome measure will be the global motor score from the motor assessment scale(MAS) testing which includes eight areas of assessment in eight areas of motor function.The MAS evaluates performance on functional tasks using a 7-point ordinal scale(0-6) in each of eight domains-moving from supine to side lying,supine to sitting over the edge of a bed, balanced sitting,moving from sitting to standing,walking,upper-arm function,hand movements(e.g., drawing a line),and advanced hand activities(e.g. combing the back of the head) rather than isolated movements. A score of 6 on each item, or an overall score of 48 indicates optimal motor behavior, and a lower score would indicate less than optimal motor behavior.

SECONDARY OUTCOMES:
Determine the correlation of periventricular tract injury in intraventricular hemorrhage(IVH) complicating intracerebral hemorrhage (ICH) with subsequent incontinence. | Ongoing/completed end of August 2020
  Determine the correlation of periventricular tract injury in IVH complicating ICH as measured by diffusion tensor imaging (DTI) with subsequent incontinence as measured by the Urogenital Distress Inventory (UDI-6),a 6 question measure of urinary continence that is highly reliable.The UDI-6 assessment scoring includes item responses that are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly."The average score of items responded to is calculated,which ranges from 0 to 3,is multiplied by 33 1/3 to put scores on a scale of 0 to 100.The lower score would indicate a better outcome and a higher score would indicate a worse outcome.
Determine the correlation of periventricular tract injury in intraventricular hemorrhage(IVH) with complicating intracerebral (ICH) with subsequent gait ataxia. | Ongoing/completed end of August 2020
  Determine the correlation of periventricular tract injury in IVH complicating intracerebral(ICH) as measured by diffusion tensor imaging(DTI) with subsequent gait ataxia as measured by motor assessment scale(MAS).The MAS includes eight areas of assessment in eight areas of motor function and evaluates performance on functional tasks using a 7 point ordinal scale(0-6) in each of the eight domains:moving from supine to side lying,supine to sitting over the edge of a bed,balanced sitting,moving from sitting to standing,walking, upper-arm function,hand movements(e.g., drawing a line), and advanced hand activities(e.g. combing the back of the head)rather than isolated movements.A score of 6 on each item,or an overall score of 48 indicates optimal motor behavior,and a lower score would indicate less than optimal motor behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Woo, MD, MS, Principal Investigator — State University of New York at Buffalo
Locations (8):
- United States (8):
  - University of Illinois Chicago, Chicago, Illinois
  - Baptist Health Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No